CLINICAL TRIAL: NCT06651632
Title: WATER IV Prostate Cancer: Aquablation Versus Radical Prostatectomy for the Treatment of Localized Prostate Cancer
Brief Title: WATER IV Prostate Cancer
Acronym: WATER IV PCa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP0005
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Cancer
Keywords: Aquablation therapy; Aquablation; Prostate cancer; AQUABEAM; radical prostatectomy; HYDROS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Aquablation Therapy (Experimental): The Aquablation Therapy arm will receive Aquablation with either the AQUABEAM Robotic System or HYDROS Robotic System
  Interventions: Device: Aquablation Therapy
- Radical Prostatectomy (Active Comparator): The radical prostatectomy arm will receive the standard of care radical prostatectomy procedure.
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Device: Aquablation Therapy — The AquaBeam Robotic System and the HYDROS Robotic System utilize high-velocity sterile saline waterjet to resect prostate tissue, guided by real-time visualization through cystoscopy and transrectal ultrasound imaging. This minimally invasive surgical procedure is called the Aquablation therapy.
  Arms: Aquablation Therapy
Procedure: Radical Prostatectomy — Radical prostatectomy is a surgery that is performed through an incision in the lower abdomen or perineum, or with a laparoscope or robotic system to remove the entire prostate gland.
  Arms: Radical Prostatectomy

SUMMARY:
This is a multicenter, prospective, randomized clinical trial that aims to assess the safety and efficacy of Aquablation Therapy in men with low-risk to intermediate to high-risk localized prostate cancer who are candidates for, or have opted for, prostatectomy. Participants will be randomized to either Aquablation Therapy or radical prostatectomy and followed up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Biological male with age ≥ 45 years at the time of consent
2. Biopsy positive Grade Group 1-3 prostate cancer
3. Are candidates for prostatectomy or, in the case of GG1 disease, have already selected a radical therapy as their treatment.
4. Clinical Stage ≤ T2c
5. PSA ≤ 20 ng/ml
6. Prostate volume ≥25 ml

Exclusion Criteria:

1. Any prior or current local or systemic treatment for prostate cancer, including but not limited to surgery, radiation therapy (external or brachytherapy), tissue ablation, hormone therapy or chemotherapy.
2. Patients with previous surgical or minimally invasive treatment of benign prostatic hyperplasia within the prior 3 months of study treatment.
3. Evidence of lymph node, bone metastasis, extracapsular extension or seminal vesicle invasion.
4. Patient is unwilling to accept a blood transfusion if required.
5. Any condition or history of illness or surgery that may pose an additional risk to patients undergoing the Aquablation or radical prostatectomy procedure such as:

5a. Medical conditions that preclude the use of anesthesia; 5b. Any condition or history of active rectal inflammatory bowel disease or other factors which might increase the risk of rectal injury (i.e. fistula formation); 5c. Patient is unable to stop anticoagulants or antiplatelet agents prior to study treatment per standard of care; 5d. Any other condition or history of infection, illness or surgery that in the opinion of the investigator might affect the outcome of the study procedure, study conduct, and study results; or pose additional risks to the patient (e.g., other cancer, active urethral stricture disease).

6. Patients who are unable to provide informed consent due to cognitive impairment, legal status (such as incarceration), or other factors limiting autonomy or unwilling or unable to follow study instructions including randomization and complete all required study visits through 10 years. This includes individuals with severe cognitive disabilities, those under legal guardianship, or those currently incarcerated.

7. Patient currently participating in other studies unless approved by Sponsor in writing.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2037-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pad use for urinary incontinence | 6 Months
Rate of erectile dysfunction | 6 Months

SECONDARY OUTCOMES:
Rate of pad use for urinary incontinence | 3 Months
Rate of erectile dysfunction | 3 Months
Stable or improved Grade Group at 1 year compared to baseline (Aquablation arm only) | 1 Year

CONTACTS AND LOCATIONS:
Locations (37):
- United States (26):
  - Arizona State Urological Institute, Chandler, Arizona
  - East Valley Urology Center, Mesa, Arizona
  - University of Southern California, Los Angeles, California
  - Boulder Medical Center, Boulder, Colorado
  - Advanced Research, Delray Beach, Florida
  - University of Miami, Miami, Florida
  - Florida Urology Partners, Tampa, Florida
  - Trophy Point Urology, Tampa, Florida
  - Georgia Urology, Atlanta, Georgia
  - Mountain View Hospital, Idaho Falls, Idaho
  - University of Chicago, Chicago, Illinois
  - Endeavor Health, Glenview, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Kansas City Urology Care, North Kansas City, Missouri
  - Kearney Urology Center, Kearney, Nebraska
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Integrated Medical Professionals, PLLC, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MUSC, Charleston, South Carolina
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Potomac Urology, Alexandria, Virginia
  - Advocate Aurora Research Institute, Sheboygan, Wisconsin
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- Universitätsklinikum OWL der Universität Bielefeld, Bielefeld, Germany
- Chinese University of Hong Kong, Shatin, Hong Kong
- Hospital Cruz Vermelha, Lisbon, Portugal
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (5):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hamsphire
  - Norfolk & Norwich University Hospital, Colney, Norwich
  - Guy's Hospital, London
  - The Royal Marsden Hospital, London
  - Royal Free Hospital, London